CLINICAL TRIAL: NCT04916067
Title: Stoma Closure and Reinforcement (SCAR)-II Trial: A Single Center Pilot Study of the Safety of a Mesh Reinforcement of Ileostomy Closure to Prevent Hernia Formation in Inflammatory Bowel Disease Patients
Brief Title: Stoma Closure and Reinforcement Trial ll
Acronym: SCAR-ll
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: terminated due to inability to complete the study
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Becton, Dickinson and Company (Industry)
Responsible Party: Principal Investigator, Matthew Z. Wilson, Assistant Professor of Surgery, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY02000875
Record Dates: First submitted 2021-06-01; First posted 2021-06-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Ileostomy - Stoma; Inflammatory Bowel Diseases
Keywords: ileostomy; hernia; inflammatory bowel disease; IBD
MeSH Terms: conditions — Inflammatory Bowel Diseases; Hernia

STUDY DESIGN:
Intervention Model Description: Modified Simon-Two Step. An initial cohort of 5 patients will be enrolled and treated sequentially with 30 day follow-up. If stopping criteria are not met, the cohort will be expanded to an additional 15 patients followed concurrently for the duration of the study period
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Intervention (Experimental): Patients undergoing mesh implantation during ileostomy closure to reinforce the abdominal wall
  Interventions: Device: Mesh Implantation

INTERVENTIONS:
Device: Mesh Implantation — Implantation of Phasix™ Soft Mesh - a knitted monofilament mesh scaffold using Poly-4-hydroxybutyrate (P4HB), a biologically derived material - to prevent hernia formation

SUMMARY:
Hernia formation at sites of ostomy closure is a common complication. The investigator believes that using evidence based hernia repair techniques as a preventive measure during closure of ostomies will reduce the incidence of hernia formation. In this trial, the investigator will pilot a novel technique of monofilament bioresorbable mesh reinforcement of the abdominal wall defects that remain after closure of an ileostomy to evaluate for safety and begin to evaluate the effectiveness compared to standard techniques.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18years.
2. Patient is undergoing closure of loop ileostomy.
3. Patient has a diagnosis of Inflammatory bowel disease treated with resection and diverting loop ileostomy.
4. Patient has been evaluated by a qualified surgeon and found to be a suitable candidate for surgery.

Exclusion Criteria:

1. Pre-existing systemic infection at the time of ileostomy takedown
2. Cirrhosis, chronic renal failure requiring dialysis, or collagen disorder
3. Previous abdominal hernia repair with mesh placement
4. Concurrent surgical procedures in addition to closure of diverting loop ileostomy
5. Ileostomy closure not completed through the previous stoma site (i.e. those requiring exploratory laparotomy for closure)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2024-08-05 (Actual)

PRIMARY OUTCOMES:
Incidence of wound occurrences | 30 days
  Incidence of wound occurrences (defined as superficial surgical site infection [s-SSI], deep surgical site infection [d-SSI], organ space surgical site infection [O-SSI], dehiscence, and seroma formation) at 30 days, with particular attention to wound occurrences requiring procedural intervention, including but not limited to, operative debridement, radiographically guided drain placement, or excision of the mesh will be assessed.

SECONDARY OUTCOMES:
Incidence of hernia formation | 30 days, 6 months
  The incidence of hernia formation at the ileostomy site on a prospective basis at 30 days and at 6 months from the date of ileostomy closure.
Quality of Life after mesh implantation | 30 days, 6 months
  Patient will be evaluated with regards to their quality of life outcomes the PROMIS SF 2.0, Ability to Participate in Social Roles and Activities, instrument at 30 days and 6 months from the date of ileostomy closure.
Bowel Function after mesh implantation | 30 days, 6 months
  Patient will be evaluated with regards to their bowel function using the Colorectal Functional Outcome (COREFO) instrument at 30 days and 6 months from the date of ileostomy closure.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Z Wilson, MD, Msc, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goldwag JL, Wilson LR, Ivatury SJ, Pauli EM, Tsapakos MJ, Wilson MZ. Stoma closure and reinforcement (SCAR): A study protocol for a pilot trial. Contemp Clin Trials Commun. 2020 Jun 9;19:100582. doi: 10.1016/j.conctc.2020.100582. eCollection 2020 Sep. PMID 32577580